CLINICAL TRIAL: NCT07146035
Title: Feasibility of a Newly Developed Ostomy Prototype
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP369
Record Dates: First submitted 2025-07-25; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Stoma - Ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigation (one armed study) (Experimental)
  Interventions: Device: CP369 Feasibility of a newly developed ostomy prototype (only one intervention)

INTERVENTIONS:
Device: CP369 Feasibility of a newly developed ostomy prototype (only one intervention) — The study is an open-label, single-arm, comparative study, investigating the feasibility of the prototype in subjects with ileostomy. The study is comparing the prototype exposed only to sweat (abdominal side) with the prototype exposed to sweat and output (peristomal side). Meaning, subjects are their own control.

SUMMARY:
Despite the development of better stoma products, individuals with intestinal stomas can experience leakage problems, which negatively affect their quality of life. To overcome this, Coloplast are in the process of developing a leakage measurement device. Each participant will undergo five 24-hour test periods over three weeks, wearing the prototype around the stoma (Test) and on the opposite side (Control).

ELIGIBILITY:
Inclusion Criteria:

Has given written informed consent Is at least 18 years old Has full legal capacity Is able (assessed by the investigator) and willing to adhere to study procedures during study duration.

Has had an ileostomy for at least 30 days. Has been self-managing their own ostomy product for at least 14 days. Has experienced leakage under the baseplate at least 3 times within the past 2 weeks.

Is able to fit one of the two test product sizes (Ø50mm or Ø60mm). Uses a flat baseplate Is willing to change their baseplate daily Has intact peristomal skin (assessed by the investigator) Is able to use a smartphone with camera

Exclusion Criteria:

Is participating in any other clinical investigation during this investigation Has previously participated or completed this investigation Has a known hypersensitivity towards the prototype used in the investigation Is pregnant Is breast feeding Has more than one ostomy synchronously Has ongoing non-healed abdominal wounds Has planned MR scans during the 24-hour test recording

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
To test the system performance of the prototype. | 3 weeks from enrollment to end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast, UserLab, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: Undecided